CLINICAL TRIAL: NCT04242017
Title: A Randomized, Multicenter, Prospective Phase II Trial to Assess the Effect of Short- Versus Long-term Adjuvant ADT With High Dose Salvage Radiotherapy on Distant Metastasis Free Survival in Patients With Biochemical Relapse After Radical Prostatectomy
Brief Title: Long-term Better Than Short-term ADT With Salvage RT
Acronym: LOBSTER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S61996
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
Keywords: pN0; biochemical recurrence; salvage radiation therapy; hormonal treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- salvage RT + 6 months ADT (Active Comparator): 70 Gy to the prostate bed (2 Gy/fraction) + 6 months ADT
  Interventions: Drug: Triptoreline
- salvage RT + 24 months ADT (Experimental): 70 Gy to the prostate bed (2 Gy/fraction) + 24 months ADT
  Interventions: Drug: Triptoreline

INTERVENTIONS:
Drug: Triptoreline — Comparison of the duration of ADT (Triptoreline)

SUMMARY:
A randomized, multicenter, prospective PHASE II trial to assess the effect of short- versus long-term adjuvant ADT with high dose salvage radiotherapy on distant metastasis free survival in case of biochemical relapse (BR) after radical prostatectomy.

DETAILED DESCRIPTION:
Radical prostatectomy (RP) is one of the standard treatment options for localized and locally advanced prostate cancer. RP should be combined with an extended pelvic lymph node dissection (ePLND) when the risk of pelvic involvement becomes substantial, at least 7%. In case of node-negative disease (pN0), adverse pathological features at examination of the RP-specimen such as extra-capsular extension (ECE), seminal vesicle invasion (SVI) and positive surgical margins (PSM) increase the risk of biochemical relapse (BR) and/or isolated local relapse (LR). Both a BR and LR, if not adequately treated, can finally result in the development of distant metastasis.

In case of BR and/or LR, salvage radiotherapy (SRT) is the only treatment option with curative intent. Several factors play a significant role in predicting the outcome after SRT: Gleason score, pre-SRT PSA, pre-SRT doubling time, SVI, SRT dose and duration of adjuvant androgen deprivation therapy (ADT) associated with SRT. The 2 latter variables have never been tested in a randomized controlled trial. The GETUG-AFU 16 trial randomized between no vs. 6 months ADT while patients received 66 Gy to the prostate bed and 46 Gy to the pelvis. Moreover, the pN0 status was not needed for inclusion. Also the RADICALS trial is currently running this comparison with a radiation dose of 66 Gy to the prostate bed and also no information on pN status is needed to be included in this study. In the LOBSTER study, the pN0 status is obligatory and the prescription dose is set at 70 Gy to the prostate bed and seminal vesicles. These conditions make this study unique compared to other already conducted and currently running trials.

In previous work, it has been demonstrated that ADT, added for 6 months to SRT, significantly improved biochemical relapse free survival at 5 years. Added to this, there is recent evidence that using a longer schedule of adjuvant ADT might be beneficial when compared to a 6-months schedule. Unfortunately, none of these suggestions are based on evidence coming from a randomized controlled trial.

Therefore, this randomized phase 2 trial 'LOBSTER' is conducted, comparing 6 versus 24 months of adjuvant ADT together with high-dose SRT in case of BR after RP in pN0 prostate cancer patients

ELIGIBILITY:
Inclusion Criteria:

* History of histologically proven prostate cancer, treated with RP and ePLND. All patients have to be pN0. The minimal template for ePLND is defined as the removal of the external iliac, internal iliac and obturator nodes (standard template). Removal of the presacral and common iliac nodes is left at the discretion of the treating urologist.
* Asymptomatic PSA-rise post-RP, defined as a value equal to or more than 0.2µg/l and at least confirmed once (interval ≥2 weeks, confirmation PSA level should be higher). In case of Gleason 8-10, pT3b or R1 resection, an asymptomatic PSA-rise post-RP starting from ≥0.15 µg/l is allowed for inclusion. If the PSA-level is less than 0.4 ng/ml, no additional staging for distant metastasis is required before inclusion in the trial. The patient will be offered the opportunity to participate in a diagnostic sub-study with investigational imaging with 18F PSMA PET CT. However in case of PSA-level >0.4 ng/ml, biological imaging using 18F-PSMA or 68Ga-PSMA is mandatory as this is not considered investigational anymore. Therefore the patient cannot anymore take part in the diagnostic sub-study and (un-blinded) PET-CT is obligatory to rule out lymph node (N) and /or distant metastasis (M1a-c) before inclusion.
* Testosterone levels within above 150 ng/dl.
* ECOG 0-1
* Life expectancy more than 5 years
* Signed informed consent

Exclusion Criteria:

* Presence of pN1 disease at original surgical specimen.
* Presence of distant metastasis at time of referral (M1a-c). If PSA more than 0.4 ng/ml, imaging with PET-CT is required to rule out distant metastasis (see above). Other additional imaging modalities (CT scan, bone scintigraphy...) are allowed but left at the discretion of the treating centre.
* Undetectable PSA (less than 0.2 ng/ml) at time of referral.
* Previous RT making new RT impossible (overlapping treatment fields).
* Known contraindications to irradiation (Ulcerative Colitis, Crohn Disease, Ataxia Teleangiectasia…)
* Active treatment with ADT or PSA modulating drugs (finasteride, dutasteride, high-dose corticoids…)
* Not able understanding treatment protocol or signing informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | 5 years
  Time to appearance of M1a-b-c disease. In order to assess the absence/presence of M1a-M1c disease as early as possible, top-of-the-line imaging will be conducted in case of BR during follow-up after SRT and after agreement of the multidisciplinary uro-oncology team. Time point zero is the last day of radiotherapy (also applies for secondary endpoints). Top of the line imaging includes: CT thorax abdomen and bone scintigraphy (standard). PSMA PET-CT is allowed but not obligatory. Patients who are also included in the diagnostic imaging study are required to receive a PSMA PET-CT. Whole body MRI is allowed but not obligatory. BR is defined as any rise in PSA above the level of 0.2 ng/ml after a postradiotherapy nadir or a continued rise in the serum PSA despite salvage treatment (3). In case a BR is not accompanied by metastatic progression, PSMA PET/CT will be repeated every 6 months or earlier in case of prostate cancer-related symptoms.

SECONDARY OUTCOMES:
Pelvic recurrence-free survival | up to 10 years after randomization
  time to appearance of local recurrence (prostate bed) and/or N1 disease (positive lymph node(s) below the aortic bifurcation) using PSMA PET/CT and triggered by biochemical relapse.
Clinical progression-free survival | up to 10 years after randomization
  time to appearance of any recurrence (local recurrence, N1 (positive lymph node(s) below the aortic bifurcation), M1a-c disease) and triggered by biochemical relapse.
(Palliative) Systemic therapy-free survival | up to 20 years (or more) after randomization
  time to the start of palliative ADT
Time to CRPC | up to 20 years (or more) after randomization
  time to biochemical and/or clinical progression at castrate testosterone levels (<50 ng/dl). Progression is defined as three consecutive PSA rises (1 week interval), of which at least 2 rises with a PSA level of > 2 ng/ml and a rise of 50% of the nadir PSA level, progression of bone lesions (2 or more new bone lesions detected on bone scan), progression of soft tissue lesions according to RECIST criteria or the appearance of one or more new visceral or soft tissue (inclusive lymph node) metastasis.
Cause-specific survival (CSS) | up to 20 years (or more) after randomization
  freedom from dying from prostate cancer (K-M statistics)
Overall survival (OS) | up to 20 years (or more) after randomization
  freedom from dying from any cause (K-M statistics)
Acute toxicity | during RT, up to three months after radiation therapy
  adverse effects according to the CTCAE version 4.0
Late toxicity | starting from more than three months after radiation therapy, up to 5 years after radiotherapy
  adverse effects according to the CTCAE version 4.0
Quality of life assessment | up to 5 years after randomization
  EORTC QLQ-C30
Quality of life assessment | up to 5 years after randomization
  EORTC QLQ-PR25
Quality of life assessment | up to 5 years after randomization
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, MD, PhD, Study Chair — UZ Leuven
Locations (3):
- Belgium (3):
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berghen C, Joniau S, Laenen A, Devos G, Rans K, Goffin K, Haustermans K, Meerleer G. Long- versus short-term androgen deprivation therapy with high-dose radiotherapy for biochemical failure after radical prostatectomy: a randomized controlled trial. Future Oncol. 2020 Sep;16(27):2035-2044. doi: 10.2217/fon-2020-0390. Epub 2020 Jul 15. PMID 32666822